





# Child Information and Assent Form Children aged 7-13 years

# The PORPOISE Study

A study to help doctors learn how to make me healthier before my varusderotational osteotomy surgery

#### Invitation

I am being invited to be part of a research study. A research study tries to find better ways to help children like me. It is up to me if I want to be in this study. No one will make me be part of the study. Even if I agree now to be part of the study, I can change my mind later. No one will be mad at me if I choose not to be part of this study.

# Why Are We Doing This Study?

I am having varus-derotational osteotomy (VDRO) surgery. This happens to other children too. This study is trying to make a nutrition plan for children having VDRO surgery. Nutrition is the foods that I eat and liquids that I drink. This study is also trying to find out if I have enough iron in my blood. Everyone has iron in their blood, but some children having VDRO surgery don't have enough iron in their blood. This study wants to find out if better nutrition and iron treatment will help patients feel better after their VDRO surgery.

# What Will Happen in This Study?

If I decide to be in this study, I will meet with a dietitian. A dietitian looks at my nutrition. A dietitian might help change my nutrition during the months before my surgery to make me healthier before I come to hospital for my surgery. I will have my blood taken twice, to see if I have enough iron in my blood. My blood will be taken after I meet with the dietitian and again before my surgery. If I don't have enough iron in my blood, I might have to take some iron pills and I might have to eat different foods, to make my nutrition better. My parents will fill out surveys, which will be sent to their emails. If my family decides to take part, we will get a \$25 Starbucks gift card.

We will also be able to do an interview while I am at the hospital if we want to. It is up to us if we want to be in the interview. If my family decides to be in the interview, we will get a second \$25 Starbucks gift card.

# Who Is Doing This Study?

Dr. Teresa Skelton and other doctors from the BC Children's Hospital will be doing this study. They will answer any questions I have about the study. I can also call them at 604-875-2711.







# Can Anything Bad Happen to Me?

If I have to take iron pills, they might make my tummy hurt and make my poops hard. The study doctors have picked a type of iron pill that is less likely to make my tummy hurt. I might also feel a poke when I get my blood taken.

# Who Will Know I Am in the Study?

Only my doctors and people involved in the study will know I am in it. When the study is finished, the doctors will write about what was learned, to help other children. This report will not say my name or that I was in the study. My parents and I do not have to tell anyone I am in the study if we do not want to.

#### When Do I Have to Decide?

I will receive a copy of this assent form.

I have as much time as I want to think about it. I can decide at any time not to take part. I can talk to my parents about my choice.

### **Assent to Participate**

My choice to participate in this study is up to me, and I can say no or decide to stop being in the study at any time.

I understand my doctors will look after me just the same, whether I decide to be in the study or not.

If I put my name at the end of this form, I agree to be in the study.

| Printed Name | <br>Signature | <br>Date |
|--------------|---------------|----------|